CLINICAL TRIAL: NCT00048971
Title: A Pharmacogenetic Case-Control Study of Severe Diarrhea and Life-Threatening Neutropenia in Patients Treated With Irinotecan, 5-Fluorouracil and Leucovorin
Brief Title: Genetic Trial to Study Diarrhea in Patients With Stage III Colon Cancer Who Are Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-60102; CALGB-60102; NCCTG-CALGB-60102; CDR0000257145 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Diarrhea; Neutropenia
Keywords: adenocarcinoma of the colon; stage III colon cancer; diarrhea; neutropenia
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Neutropenia; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients undergo collection of blood specimens for polymerase chain reaction and restriction fragment length polymorphism analysis. Genotyping assays are performed to determine UGT1A1 promoter genotyping, UGT1A1 coding polymorphisms, TS promoter polymorphisms, and MTHFR polymorphisms.
  Interventions: Genetic: mutation analysis; Genetic: polymorphic microsatellite marker analysis

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymorphic microsatellite marker analysis

SUMMARY:
RATIONALE: Genetic testing may help predict how patients will respond to chemotherapy drugs and may help doctors plan more effective treatment with fewer side effects.

PURPOSE: Genetic study to determine how genes affect the severity of diarrhea in patients with stage III colon cancer who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the presence of a 7 allele at the UGT1A1 locus is associated with either grade 3-4 diarrhea or grade 4 neutropenia in patients with stage III colon cancer after treatment with irinotecan, fluorouracil, and leucovorin calcium.
* Determine whether polymorphisms in the TS enhancer and/or MTHFR gene are associated with grade 3-4 diarrhea in these patients after treatment with fluorouracil and leucovorin calcium.
* Determine whether polymorphisms in UGT1A1, TS, MTHFR, CYP3A4, or CYP3A5 are associated with either grade 3-4 diarrhea or grade 4 neutropenia in these patients after treatment with irinotecan, fluorouracil, and leucovorin calcium.

OUTLINE: Patients are stratified according to prior therapy (irinotecan, fluorouracil, and leucovorin calcium vs fluorouracil and leucovorin calcium) and prior toxic effects (grade 3-4 diarrhea vs grade 4 neutropenia vs grade 1 or lower diarrhea AND grade 2 or lower neutropenia).

Patients undergo collection of blood specimens for polymerase chain reaction and restriction fragment length polymorphism analysis. Genotyping assays are performed to determine UGT1A1 promoter genotyping, UGT1A1 coding polymorphisms, TS promoter polymorphisms, and MTHFR polymorphisms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III adenocarcinoma of the colon
* Enrolled on CALGB-89803 and must fall into 1 of the following categories:

  * Received irinotecan, fluorouracil, and leucovorin calcium and experienced at least 1 of the following:

    * Grade 3-4 diarrhea
    * Grade 4 neutropenia
    * Grade 1 or lower diarrhea AND grade 2 or lower neutropenia
  * Received fluorouracil and leucovorin calcium and experienced at least 1 of the following:

    * Grade 3-4 diarrhea
    * Grade 1 or lower diarrhea AND grade 2 or lower neutropenia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with adenocarcinoma of the colon and previously enrolled on CALGB-89803.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2002-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
response | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark J. Ratain, MD, Study Chair — University of Chicago
Locations (84):
- United States (82):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center of Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dalas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- McGill University, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico, Puerto Rico